CLINICAL TRIAL: NCT02576353
Title: A Phase 1, Open-label, Randomized, Single Ascending Dose Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Fentanyl Sublingual Spray and Fentanyl Citrate Intravenous (IV) in Opioid Naive Subjects
Brief Title: Fentanyl Sublingual Spray and Fentanyl Citrate Intravenous (IV) in Opioid Naive Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: INSYS Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: INS002-15-049
Record Dates: First submitted 2015-10-13; First posted 2015-10-15 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Pharmacokinetics and Pharmacodynamics
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 (Experimental): After a 10-hour fast, the 10 participants in this cohort are randomized to receive Fentanyl Sublingual (under the tongue) Spray (FSS) 100 mcg (n=8), or Fentanyl Citrate Intravenously (FCIV) 50 mcg (n=2).
  Interventions: Drug: Fentanyl; Drug: Fentanyl Citrate
- Cohort 2 (Experimental): After a 10-hour fast, the 10 participants in this cohort are randomized to receive FSS 200 mcg (n=8), or FCIV 50 mcg (n=2).
  Interventions: Drug: Fentanyl; Drug: Fentanyl Citrate
- Cohort 3 (Experimental): After a 10-hour fast, the 10 participants in this cohort are randomized to receive FSS 400 mcg (n=8), or FCIV 50 mcg (n=2).
  Interventions: Drug: Fentanyl; Drug: Fentanyl Citrate
- Cohort 4 (Experimental): After a 10-hour fast, the 10 participants in this cohort are randomized to receive FSS 600 mcg (n=8), or FCIV 50 mcg (n=2).
  Interventions: Drug: Fentanyl; Drug: Fentanyl Citrate
- Cohort 5 (Experimental): After a 10-hour fast, the 10 participants in this cohort are randomized to receive FSS 800 mcg (n=8), or FCIV 50 mcg (n=2).
  Interventions: Drug: Fentanyl; Drug: Fentanyl Citrate

INTERVENTIONS:
Drug: Fentanyl — Fentanyl Sublingual Spray (FSS)
Drug: Fentanyl Citrate — Fentanyl Citrate IV (FCIV)

SUMMARY:
The primary objective of this study is to determine the pharmacokinetic and pharmacodynamic relationship of a single dose of fentanyl sublingual spray in opioid naive subjects. The secondary objective is to determine the safety and tolerability of fentanyl sublingual spray in opioid naive subjects.

ELIGIBILITY:
Inclusion Criteria:

* Meets protocol-specified criteria for qualification and contraception
* Willing and able to remain confined in the study unit for the entire duration of each treatment period and comply with restrictions related food, drink and medications
* Voluntarily consents to participate and provides written informed consent prior to any protocol-specific procedures

Exclusion Criteria:

* History or current use of over-the-counter medications, dietary supplements, or drugs (including nicotine and alcohol) outside protocol-specified parameters
* Signs, symptoms or history of any condition that, per protocol or in the opinion of the investigator, might compromise:

  1. the safety or well-being of the participant or study staff
  2. the safety or well-being of the participant's offspring (such as through pregnancy or breast-feeding)
  3. the analysis of results

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Maximum concentration | 0 (pre-dose), 5, 10, 20, 30 and 40 minutes after dosing and at 1, 1.25, 1.5, 2, 4, 6, 8, 10, 12, 16, and 24 hours after dosing
Time to maximum concentration | 0 (pre-dose), 5, 10, 20, 30 and 40 minutes after dosing and at 1, 1.25, 1.5, 2, 4, 6, 8, 10, 12, 16, and 24 hours after dosing
Area under the plasma concentration-time curve from 0 to the final time with a concentration at or above the limit of quantitation (LoQ) | 0 (pre-dose), 5, 10, 20, 30 and 40 minutes after dosing and at 1, 1.25, 1.5, 2, 4, 6, 8, 10, 12, 16, and 24 hours after dosing
Area under the plasma concentration-time curve from 0 to infinity | 0 (pre-dose), 5, 10, 20, 30 and 40 minutes after dosing and at 1, 1.25, 1.5, 2, 4, 6, 8, 10, 12, 16, and 24 hours after dosing
Apparent elimination rate constant in the terminal phase by noncompartmental analysis | 0 (pre-dose), 5, 10, 20, 30 and 40 minutes after dosing and at 1, 1.25, 1.5, 2, 4, 6, 8, 10, 12, 16, and 24 hours after dosing
Elimination half-life | 0 (pre-dose), 5, 10, 20, 30 and 40 minutes after dosing and at 1, 1.25, 1.5, 2, 4, 6, 8, 10, 12, 16, and 24 hours after dosing
Apparent oral clearance of drug following extravascular administration | 0 (pre-dose), 5, 10, 20, 30 and 40 minutes after dosing and at 1, 1.25, 1.5, 2, 4, 6, 8, 10, 12, 16, and 24 hours after dosing
Volume of distribution during terminal phase following extravascular administration | 0 (pre-dose), 5, 10, 20, 30 and 40 minutes after dosing and at 1, 1.25, 1.5, 2, 4, 6, 8, 10, 12, 16, and 24 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Neha N Parikh, Study Director — INSYS Therapeutics Inc
Locations (1):
- Lotus Clinical Research, Pasadena, California, United States

REFERENCES:
- [Derived] Rauck R, Oh DA, Parikh N, Koch C, Singla N, Yu J, Nalamachu S, Vetticaden S. Pharmacokinetics and safety of fentanyl sublingual spray and fentanyl citrate intravenous: a single ascending dose study in opioid-naive healthy volunteers. Curr Med Res Opin. 2017 Nov;33(11):1915-1920. doi: 10.1080/03007995.2017.1352496. Epub 2017 Aug 11. PMID 28681626